CLINICAL TRIAL: NCT06185985
Title: A Phase IV, Open-Label, Decentralized Clinical Trial to Evaluate the Efficacy and Safety of Qelbree® in Adults With Attention-Deficit/Hyperactivity Disorder and Mood Symptoms
Brief Title: Open-label Safety and Efficacy of SPN-812 (Viloxazine Extended-release Capsule) in Adults With ADHD and Mood Symptoms
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812P413
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label Treatment (Experimental): SPN-812 (200mg to 600mg once daily) for up to 14 weeks
  Interventions: Drug: SPN-812

INTERVENTIONS:
Drug: SPN-812 — SPN-812 (200mg to 600mg once daily)
  Other Names: viloxazine extended-release capsules; Qelbree

SUMMARY:
Open label, flexible dose, decentralized clinical trial evaluating the efficacy and safety of SPN-812 in adults with ADHD and mood symptoms.

DETAILED DESCRIPTION:
This is a Phase IV, open-label, flexible dose, decentralized clinical trial to evaluate the efficacy and safety of SPN-812 in adults with ADHD and mood symptoms. Adults 18 years and older with ADHD will be recruited, consented and screened for eligibility. Following the Screening Period (up to 4 weeks), eligible participants will be treated with Study medication for up to 14 weeks (Treatment Period). The total study duration is approximately 18 weeks, and there are up to 6 virtual study visits (or Televisits). All Televisits are conducted via an application downloaded to participant's mobile phone. There are up to 2 Televisits during the Screening period and 3 Televisits during the Treatment period. Subjects initiate SPN-812 dosing at 200 mg once daily during first week, and then titrate up to 400mg once daily during the second week. At the Investigator's discretion, based subject's clinical response and tolerability, the dose of SPN-812 can be increased or decreased to optimal dose within the range between 200 and 600 mg once daily during the remaining Treatment period. Participants will answer questions during structured clinical interviews with an investigator during Televisits and complete additional questionnaires and scales via the mobile app.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, a participant must meet all of the following criteria:

1. Is male or female, ≥18 years of age.
2. Is willing and capable of providing and signing electronic informed consent.
3. Has a primary diagnosis of ADHD based on the Diagnostic and Statistical Manual of Mental Disorders; Fifth Edition, Text Revision (DSM-5-TR) as confirmed with the Mini-International Neuropsychiatric Interview for ADHD Studies (MINI-AS).
4. Has an AISRS Total score ≥24 at Screening.
5. Has a CGI-S score ≥3 at Screening.
6. Has a MADRS (SIGMA) Total score >22 at Screening and/or HAM-A (SIGH-A) Total score >22 at Screening.
7. If potential participant is a biological female, one of the following (a, b, or c) must be met:

   1. Has undergone menopause, defined as a biological female who reports amenorrhea for at least 12 consecutive months prior to providing informed consent.
   2. Is a non-pregnant Female of Childbearing Potential (FOCP) who is not seeking fertility treatment during the study and agrees to use one of the following acceptable birth control methods beginning 14 days prior to the first dose of study medication, throughout the study while taking study medication, and for 7 days following the last dose of study medication: i. Hormonal contraceptive; ii.Barrier method: simultaneous use of male condom and diaphragm or cervical cap with spermicidal foam/gel/film/cream/suppository.
   3. Has had bilateral tubal ligation, hysterectomy, bilateral oophorectomy (permanently sterilized) at least 6 months prior to providing informed consent.
8. If potential participant is a biological male, one of the following must be met:

   1. Is capable of having children and agrees to use 2 methods of contraception beginning 14 days prior to the first dose of study medication, throughout the study while taking study medication, and for 7 days following the last dose of study medication.
   2. Has had sterilization surgery (permanently sterilized) at least 6 months prior to providing informed consent.
9. Owns a functioning smartphone device, has access to an internet connection (Wi-Fi or data plan), is willing to download and use the study mobile app throughout the study, and is willing to have visual telemedicine appointments (televisits) at times designated in the study protocol.

Exclusion Criteria:

A participant who meets any of the following criteria will be excluded from participation in the study:

1. Has a history of substance use disorder (alcohol, opioids, etc.) within the last 6 months prior to providing informed consent with exception of nicotine and cannabis.
2. Is currently taking or has taken Qelbree for treatment of ADHD in the last 3 months or is currently taking another non-stimulant medication for treatment of ADHD, like atomoxetine (Strattera), Clonidine (Catapres, Kapvay) or Guanfacine (Tenex, Intuniv). Stimulant medications for ADHD and most medications for mood symptoms (symptoms of depression and/or anxiety) are allowed.
3. Is taking a prohibited concomitant medication per the Qelbree prescribing information.
4. Is a FOCP who is pregnant, nursing, sexually active with a male partner and not willing to use one of the acceptable birth control methods throughout the study and/or is seeking fertility treatment.
5. Has a history of moderate or severe head trauma or other neurological disorder or systemic medical disease that, in the Investigator's opinion, is likely to affect central nervous system functioning. This would include participants with:

   1. A current diagnosis of a major neurological disorder; or
   2. Seizures, seizure disorder or seizure-like events; or a history of seizure disorder within the immediate family (siblings, parents); or
   3. Encephalopathy
6. Has attempted suicide within the 6 months prior to the C-SSRS assessment at Screening, or is at significant risk of suicide, either in the opinion of the Investigator or defined as a "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior on the C-SSRS within the 6 months prior to the C-SSRS assessment at Screening.
7. Is currently participating in another clinical trial or has participated in a clinical trial within the 60 days prior to providing informed consent.
8. Has any history of schizophrenia, schizoaffective disorder, or bipolar disorder, or has any other psychiatric disorders in the investigator's clinical judgement would interfere with their ability to participate in the study.
9. Has any unstable, clinically significant cardiovascular condition that in the investigator's clinical judgement would preclude their participating in the study.
10. Has any disease or taking any medication that could, in the Investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with study conduct or interpretation of results.
11. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeat or palpitations or near drowning with hospital admission.
12. In the Investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Adult ADHD Investigator Symptom Rating Scale (AISRS) Total score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Investigator Symptom Rating Scale (AISRS) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the ratings of all 18 items yields the raw Total score (range: 0-54; the higher the Total score, the more severe the ADHD symptoms). Post-baseline raw Total scores are converted to a change from baseline Total score. A lower change from baseline Total Score (<0) represents a better outcome.

SECONDARY OUTCOMES:
Change from baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) Inattention Subscale score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Investigator Symptom Rating Scale (AISRS) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the ratings of the 9 IA items yields the raw IA subscale score (range: 0-27; the higher the IA Subscale score, the more severe the IA symptoms). Post-baseline raw Subscale score is converted to a change from baseline Subscale score. A lower change from baseline Subscale Score (<0) represents a better outcome.
Change from baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) Hyperactivity/Impulsivity Subscale score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Investigator Symptom Rating Scale (AISRS) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the ratings of the 9 HI items yields the raw HI subscale score (range: 0-27; the higher the HI Subscale score, the more severe the HI symptoms). Post-baseline raw Subscale score is converted to a change from baseline Subscale score. A lower change from baseline Subscale Score (<0) represents a better outcome.

OTHER OUTCOMES:
Change from baseline in Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) Total score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) is an ADHD-specific rating scale designed and validated to assess self-ratings of current ADHD symptomatology in adults. The ASRSv1.1-SC consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The subject rates the frequency of each item on a 5-point scale, where 0=never, 1=rarely, 2=sometimes, 3=often, and 4=very often. The sum of the ratings of all 18 items yields the raw Total score (range: 0-72; the higher the Total score, the more severe the ADHD symptoms). Post-baseline raw Total scores are converted to a change from baseline Total score. A lower change from baseline Total Score (<0) represents a better outcome.
Change from baseline in the Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) Inattention Subscale score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) is an ADHD-specific rating scale designed and validated to assess self-ratings of current ADHD symptomatology in adults. The ASRSv1.1-SC consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The subject rates the frequency of each item on a 5-point scale, where 0=never, 1=rarely, 2=sometimes, and 3=often, and 4=very often. The sum of the ratings of the 9 IA items yields the raw IA subscale score (range: 0-36; the higher the IA Subscale score, the more severe the IA symptoms). Post-baseline raw Subscale score is converted to a change from baseline Subscale score. A lower change from baseline Subscale Score (<0) represents a better outcome.
Change from baseline in the Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) Hyperactivity/Impulsivity Subscale score by visit. | Baseline and Week 4, 9, and 14
  The Adult ADHD Self-Report Scale (v1.1) Symptoms Checklist (ASRSv1.1-SC) is an ADHD-specific rating scale designed and validated to assess self-ratings of current ADHD symptomatology in adults. The ASRSv1.1-SC consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (IA; 9 items) and Hyperactivity/Impulsivity (HI; 9 items). The subject rates the frequency of each item on a 5-point scale, where 0=never, 1=rarely, 2=sometimes, and 3=often, and 4=very often. The sum of the ratings of the 9 HI items yields the raw HI subscale score (range: 0-36; the higher the HI Subscale score, the more severe the HI symptoms). Post-baseline raw Subscale score is converted to a change from baseline Subscale score. A lower change from baseline Subscale Score (<0) represents a better outcome.
Change from baseline in the Clinical Global Impression of Severity (CGI-S) score by visit | Baseline and Week 4, 9, and 14
  The Clinical Global Impression of Severity (CGI-S) scale is a single item clinician-rated assessment of the severity of subject's condition (ADHD symptoms) in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated on a 7-point scale with 1 = Asymptomatic, no symptoms; 2 = Borderline, 3 = Mild, 4 = Moderate, 5 = Marked, 6 = Severe, and 7 = Among the most extreme (the higher the score, the more severe the symptoms). Post-baseline (raw) CGI-S scores are converted to a change from baseline score. A lower change from baseline CGI-S score (<0) represents a better outcome.
The Clinical Global Impression of Change (CGI-C) score by visit | Week 4, 9, and 14
  The Clinical Global Impression of Change (CGI-C) scale is a single item clinician-rated assessment of how much the subject's condition (ADHD) has improved, worsened or has not changed relative to his/her baseline state prior to the beginning of treatment. The CGI-C is rated on a 7-point scale from 1 to 7, where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse", 6 = "much worse", and 7 = "very much worse". A CGI-C score <4 represents a better outcome.
Change from baseline in the Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score at Week 14/End of Study | Baseline and Week 14
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item investigator-rated diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders and is designed to be sensitive to changes elicited by treatment. A Structured Interview Guide for the MADRS (SIGMA) was developed to improve inter- and intra-rater consistency and improve reliability. The clinician rates each of the 10 items (symptoms) on a 7-point scale [0-6 continuum, where 0=no abnormality to 6=severe]. The sum of the ratings of all 10 items yields the raw Total score (range: 0-60; the higher the Total score, the more severe the depression symptoms). The post-baseline raw Total score is converted to a change from baseline Total score. A lower change from baseline Total Score (<0) represents a better outcome.
Change from baseline in Patient Health Questionnaire 8-item (PHQ-8) Total Score by visit | Baseline and Week 4, 9, and 14
  The Patient Health Questionnaire 8-item (PHQ-8) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression per diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders. The PHQ-8 has been validated as a diagnostic and severity measure for depressive disorders in large clinical studies. The patient rates each item on 4-point scale (0-3), where 0 = not at all; 1 = several days; 2 = more than half the days; and 3 = nearly every day). The sum of the ratings of all 8 items yields the raw Total score (range: 0-24; the higher the Total score, the more severe the depression symptoms). The post-baseline raw Total score is converted to a change from baseline Total score. A lower change from baseline Total Score (<0) represents a better outcome.
Change from baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Week 14 | Baseline and Week 14
  The Hamilton Anxiety Scale (HAM-A) is a 14-item investigator-rated scale developed to assess/measure the severity of an individual's anxiety. The HAM-A has been used to assess severity of anxiety in children, adolescents, and adults in both clinical and research settings. A Structured Interview Guide for the HAM-A (SIGH-A) was developed to improve inter- and intra-rater consistency and improve reliability. The clinician rates each of the 14 items on a 5-point scale (0-4), where 0 = Not present, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very severe. The sum of the ratings of all 14 items yields the raw Total score (range: 0-56; the higher the Total score, the more severe the symptoms of anxiety). The post-baseline raw Total score is converted to a change from baseline Total score. A lower change from baseline Total Score (<0) represents a better outcome.
Change from baseline in General Anxiety Disorder 7-item (GAD-7) Total Score by visit | Baseline and Week 4, 9, and 14
  The Generalized Anxiety Disorder 7-Item (GAD-7) is a self-reported 7-item questionnaire for screening and measuring the severity of generalized anxiety disorder. The subject rates each item on 4-point scale (0-3), where 0 = "Not at all", 1 = "Several days", 2 = "Over half the days", and 3 = "Nearly every day". The sum of the 7 items yields a raw GAD-7 Total score (range between 0 to 21); the higher the Total score, the more severe the symptoms of anxiety. Post-baseline raw Total scores are converted to a change from baseline Total score. A lower change from baseline Total score (<0) represents a better outcome.
Change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Global Executive Composite (GEC) T-score at Week 14 (End of Study) | Baseline and Week 14
  The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a 75-item self-rating scale that assesses overall functioning (GEC) and 9 non-overlapping scales among 2 summary index scales (Metacognition Index [MI] and Behavioral Regulation Index [BRI]) that assess aspects of executive function and problems with self-regulation from the perspective of the individual. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 70 items yields the GEC raw score (range: 70-210), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). The post-baseline GEC T-score is converted to a change from baseline T-score. A lower change from baseline GEC T-score (<0) represents a better outcome.
Change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Behavioral Regulation Index (BRI) T-score at Week 14 (End of Study) | Baseline and Week 14
  The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales, the Metacognition Index (MI) and the Behavioral Regulation Index (BRI). The BRI captures the ability to maintain appropriate regulatory control of one's own behavior and emotional responses. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 30 items yields the BRI raw score (range: 30-90), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). The post-baseline BRI T-score is converted to a change from baseline T-score. A lower change from baseline BRI T-score (<0) represents a better outcome.
Change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Metacognition Index (MI) T-score at Week 14 (End of Study) | Baseline and Week 14
  The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales, the Metacognition Index (MI) and the Behavioral Regulation Index (BRI). MI reflects individual's ability to problem solve (includes initiate activity, generate ideas, sustain working memory, plan/organize approaches, monitor success/failure, and organize materials/environment). Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 40 items yields the MI raw score (range: 40-120), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). The post-baseline MI T-score is converted to a change from baseline T-score. A lower change from baseline MI T-score (<0) represents a better outcome.
Change from baseline in the Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Absenteeism percentage by visit | Baseline and Week 4, 9, and 14
  The Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Questionnaire is a self-assessment questionnaire that measures the impact of health problems on work productivity and regular activities based on specific health problem (e.g., ADHD). The WPAI:SHP consists of 6 questions that ask about the number of hours missed from work or regular activities due to the specific health problem. The WPAI:SHP yields 4 scores: absenteeism (percentage of time absent from work), presenteeism (percentage of time impaired/unproductive at work), total work productivity impairment (absenteeism plus presenteeism), and total activity impairment (percentage of time affected outside the workplace); range 0-100%; the higher percentage, the greater the impairment). Post-baseline percentages are converted to a change from baseline percentage. A lower change from baseline Absenteeism percentage (<0) represents a better outcome.
Change from baseline in the Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP Presenteeism percentage by visit | Baseline and Week 4, 9, and 14
  The Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Questionnaire is a self-assessment questionnaire that measures the impact of health problems on work productivity and regular activities based on specific health problem (e.g., ADHD). The WPAI:SHP consists of 6 questions that ask about the number of hours missed from work or regular activities due to the specific health problem. The WPAI:SHP yields 4 scores: absenteeism (percentage of time absent from work), presenteeism (percentage of time impaired/unproductive at work), total work productivity impairment (absenteeism plus presenteeism), and total activity impairment (percentage of time affected outside the workplace); range 0-100%; the higher percentage, the greater the impairment). Post-baseline percentages are converted to a change from baseline percentage. A lower change from baseline Presenteeism percentage (<0) represents a better outcome.
Change from baseline in the Change from baseline in the Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Work Productivity percentage by visit | Baseline and Week 4, 9, and 14
  The Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Questionnaire is a self-assessment questionnaire that measures the impact of health problems on work productivity and regular activities based on specific health problem (e.g., ADHD). The WPAI:SHP consists of 6 questions that ask about the number of hours missed from work or regular activities due to the specific health problem. The WPAI:SHP yields 4 scores: absenteeism (percentage of time absent from work), presenteeism (percentage of time impaired/unproductive at work), total work productivity impairment (absenteeism plus presenteeism), and total activity impairment (percentage of time affected outside the workplace); range 0-100%; the higher percentage, the greater the impairment). Post-baseline percentages are converted to a change from baseline percentage. A lower change from baseline Work Productivity percentage (<0) represents a better outcome.
Change from baseline in the Change from baseline in the Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Regular Activity percentage by visit | Baseline and Week 4, 9, and 14
  The Work Productivity and Activity Impairment:Specific Health Problem (WPAI:SHP) Questionnaire is a self-assessment questionnaire that measures the impact of health problems on work productivity and regular activities based on specific health problem (e.g., ADHD). The WPAI:SHP consists of 6 questions that ask about the number of hours missed from work or regular activities due to the specific health problem. The WPAI:SHP yields 4 scores: absenteeism (percentage of time absent from work), presenteeism (percentage of time impaired/unproductive at work), total work productivity impairment (absenteeism plus presenteeism), and total activity impairment (percentage of time affected outside the workplace); range 0-100%; the higher percentage, the greater the impairment). Post-baseline percentages are converted to a change from baseline percentage. A lower change from baseline Regular Activity percentage (<0) represents a better outcome.
Change from baseline in the Pittsburgh Sleep Quality Index (PSQI) Global score at Week 14 (End of Study) | Baseline and Week 14
  The Pittsburgh Sleep Quality Index (PSQI) is a validated and effective instrument used to measure the quality and patterns of sleep in adults. The PSQI is a self-rated, 19-item questionnaire out of which generate 7 component scores (or domains): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored on a 4-point scale based on an individual algorithm; range: 0 to 3, whereby 0=better and 3=worse). The sum of all 7 component scores yields the Global score (range:0 to 21); a global score >5 is associated with poor sleep quality. A post-baseline raw Global score is converted to a change from baseline Global score. A lower change from baseline Global score (<0) represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- ObvioHealth, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No